CLINICAL TRIAL: NCT03507504
Title: REspectful CAring for the AGitated Elderly. How to Best Meet the Needs of People With Dementia With Severe Behavioural Disturbances. Toward a Respectful and Cost-effective Model
Brief Title: REspectful CAring for the AGitated Elderly
Acronym: RECAGE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Europea di Ricerca Biomedica Ferb Onlus (Other)
Collaborators: Mediolanum Cardio Research (Other)
Responsible Party: Principal Investigator, Carlo Alberto Defanti, Study Coordinator, Fondazione Europea di Ricerca Biomedica Ferb Onlus
Other Study IDs: H2020 Proposal, number: 779237
Record Dates: First submitted 2018-04-09; First posted 2018-04-25 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Dementia
Keywords: psychiatric aspects
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- care pathway with SCU-B: 250 patients with dementia and behavioural and psychological symptoms of dementia (BPSD) followed up by six clinical centres with a Special Care Unit for BPSD (SCU-B)
  Interventions: Other: SCU-B
- care pathway without SCU-B: 250 patients with dementia and BPSD followed up by six clinical centres without SCU-B

INTERVENTIONS:
Other: SCU-B — SCU-B is "a residential medical structure lying outside of a nursing home, in a general hospital or elsewhere, e.g. in a private hospital, where patients with BPSD are temporarily admitted when their behavioural disturbances are not amenable to control at home".
  Groups: care pathway with SCU-B

SUMMARY:
The treatment of Behavioural and Psychological Symptoms of Dementia (BPSD) continue to raise difficult problems. Both the pharmacologic and non-pharmacologic therapies often fail to achieve the expected results. The aim of this study is to assess the short- and long-term efficacy of an intervention, the Special Care Unit for patients with BPSD (SCU-B), already implemented in some countries but not validated so far, as well as its cost-effectiveness

DETAILED DESCRIPTION:
Two cohorts of 250 patients each will be recruited by six clinical centres endowed with a SCU-B (one cohort) and six centres lacking this structure. The follow-up will last 3 years, during which patients will be visited every 6 months and submitted to a battery exploring the severity of the BPSD and the quality of life. All adverse events will be registered, as well as some anticipated occurrences (admissions to the general hospital for intercurrent diseases, admissions to a SCU-B pertaining to the clinical participating centre and, if any, admissions to a SCU-B not pertaining to the Consortium member, nursing home placement).

At the same time the quality of life of the primary caregivers will be measured, as well as their attitude toward dementia.

A cost-effectiveness analysis will be performed comparing the cohorts. Finally the time to the nursing home placement will be recorded and compared between the two cohorts

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of primary dementia (DSM IV)
* MMSE score ≤ 24
* NPI global score ≥ 32/144
* a caregiver (informal/family member or formal caregiver) who commits her/himself to accompany the patient along the three-year course of the study
* living at home (nursing home residents are excluded).

Exclusion Criteria:

* presence of uncontrolled medical disease potentially contributing to the cognitive decline and BPSD
* concomitant psychiatric disorders or chronic alcoholism
* concomitant diseases severe enough to reduce life expectancy < 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population studied is made by the outpatients with dementia referred to the memory clinics of 12 clinical centres located in seven European countries (Italy, Germany, France, Belgium, Greece, Switzerland, Norway)
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-04-19 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
change of BPSD | baseline, 6, 12, 18, 24, 30, 36 months
  Neuropsychiatric Inventory (NPI), range 0-144

SECONDARY OUTCOMES:
quality of life of patients | baseline, 6, 12,18, 24, 30, 36 months
  Quality of Life Alzheimer's Disease (QoL-AD), range 0-52
quality of life of caregivers | baseline, 6, 12, 18, 24, 30, 36 months
  Caregiver Burden Inventory (CBI), range 0-96
cost-effectiveness of SCU-B | baseline, 6, 12, 18, 24, 30, 36 months
  Resource Utilisation in Dementia (RUD)

OTHER OUTCOMES:
delayed institutionalisation | until 3 years
  Time to nursing home placement

CONTACTS AND LOCATIONS:
Overall Officials: Carlo A Defanti, M.D., Study Director — Fondazione Europea di Ricerca Biomedica
Locations (12):
- Centre Hospitalier Universitaire St Pierre, Brussels, Belgium
- Assistance Publique - Hopitaux de Paris, Paris, France
- Germany (2):
  - Zentralinstitut für Seelische Gesundheit, Mannheim, Baden-Wurttenberg
  - Charité - Universitätsmedizin Berlin, Berlin
- Aristotelio Panepistimio Thessalonikis (Greece), Thessaloniki, Greece
- Italy (5):
  - Cliniche Gavazzeni SpA, Bergamo, BG
  - Fondazione Europea di Ricerca Biomedica, Gazzaniga, BG
  - Azienda Socio Sanitaria Territoriale di Mantova, Mantova, MN
  - Azienda Unità Sanitaria Locale di Modena, Modena, MO
  - Università degli Studi di Perugia, Perugia, PG
- Sykehuset Innlandet, Ottestad, Norway
- Université de Genève, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data both for primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available six months after study completion
Access Criteria: Data access requests will be reviewed by an independent Data Safety Monitoring Board

REFERENCES:
- [Background] Koskas P, Belqadi S, Mazouzi S, Daraux J, Drunat O. [Behavioral and psychological symptoms of dementia in a pilot psychogeriatric unit: management and outcomes]. Rev Neurol (Paris). 2011 Mar;167(3):254-9. doi: 10.1016/j.neurol.2010.07.030. Epub 2010 Oct 14. French. PMID 20947112
- [Background] Delphin-Combe F, Roubaud C, Martin-Gaujard G, Fortin ME, Rouch I, Krolak-Salmon P. [Effectiveness of a cognitive-behavioral unit on behavioral and psychological symptoms of dementia]. Rev Neurol (Paris). 2013 Jun-Jul;169(6-7):490-4. doi: 10.1016/j.neurol.2012.10.017. Epub 2013 Mar 21. French. PMID 23523558
- [Background] Bianchetti A, Benvenuti P, Ghisla KM, Frisoni GB, Trabucchi M. An Italian model of dementia special care unit: results of a pilot study. Alzheimer Dis Assoc Disord. 1997 Mar;11(1):53-6. doi: 10.1097/00002093-199703000-00009. PMID 9071445
- [Derived] Cesana BM, Bergh S, Ciccone A, Cognat E, Fabbo A, Fascendini S, Frisoni GB, Froelich L, Handels R, Jori MC, Mecocci P, Merlo P, Peters O, Tsolaki M, Defanti CA. Predictors of Nursing Home Placement in a Cohort of European People with Alzheimer's Disease and Other Dementia Cases Enrolled in SCU-B or Non SCU-B Centers: The RECage Study. J Alzheimers Dis. 2024;98(3):1043-1052. doi: 10.3233/JAD-230878. PMID 38489173